CLINICAL TRIAL: NCT02046343
Title: ENLACE: A Promotora-Led Physical Activity Intervention Trial for Latinas in Texas
Brief Title: Promotora-Led Physical Activity Intervention Trial for Latinas in Texas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of South Carolina (Other); The University of Texas Health Science Center, Houston (Other); Texas A&M University (Other); Texas Tech University Health Sciences Center, El Paso (Other); University of Maryland (Other)
Responsible Party: Principal Investigator, Deborah Parra-Medina, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSC20110460H; R01HL111718 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Physical Activity
Keywords: physical activity; prevention; health disparities; behavior; community based intervention
MeSH Terms: conditions — Motor Activity; Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Experimental): Weekly promotora-led group sessions on physical activity (16 weeks) and followed by monthly telephone counseling and newsletters during the 24 week maintenance period. Promotoras will also implement environmental change strategies to increase the number of PA program offerings available to study participants.
  Interventions: Behavioral: Health education; Behavioral: Telephone Counseling; Other: Newsletter; Other: Environmental Change
- Community Health and Safety (Placebo Comparator): Weekly promotora-led group sessions on home safety/first aid (16 weeks) followed by and monthly generic health education materials and informational telephone calls during the 24 week maintenance period.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — Group health education sessions delivered by a promotora approximately 90 minutes in length. In the PA arm, health education incorporates at least 30 minutes group exercise.
Behavioral: Telephone Counseling — Brief (10 minute) telephone counseling calls delivered by promotoras using motivational interviewing techniques. The counseling calls will emphasize behavior change strategies, including self-monitoring, goal setting, reinforcement, problem solving, stimulus control, and enlisting social support.
  Arms: Physical Activity
Other: Newsletter — Educational, motivational and informational newsletters tailored for each community and hand-delivered by promotoras to participant homes.
  Arms: Physical Activity
Other: Environmental Change — Create a site atmosphere that promotes PA and increases the number of PA program offerings.
  Arms: Physical Activity

SUMMARY:
The purpose of this study it to determine if a promotora-led intervention that takes a comprehensive, multi-level, community-based approach to promoting physical activity (PA) is effective among a particularly underserved segment of Latinas. We hypothesize that Latinas in the promotora-led PA Intervention will significantly increase minutes per week of moderate-to-vigorous physical activity (MVPA) compared to Latinas in the attention-control group.

ELIGIBILITY:
Inclusion Criteria:

* women ages 18-64 years
* self-identify as Hispanic
* have a personal telephone
* reside within and intend to stay in the specified areas over the entire study period
* understand Spanish
* do not currently meet national PA recommendations

Exclusion Criteria:

* currently pregnant or plan to become pregnant
* insulin dependent diabetic
* uncontrolled hypertension
* undergoing therapy for life-threatening illnesses (chemotherapy or radiation therapy)
* positive (risk) responses on the PA Readiness Questionnaire (PAR-Q) and subsequent physician disapproval

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 712 (Actual)
Dates: Start 2012-08; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Moderate-to-vigorous physical activity (MVPA) | 16 weeks
  Minutes per week of MVPA is assessed a baseline and immediate post-intervention (16 weeks) using accelerometry. The primary outcome is the amount of change between baseline and immediate post-intervention.

SECONDARY OUTCOMES:
Change from baseline in Physical Fitness | 16 weeks
  The "2-minute step in place" test will be used to assess the amount of change in cardiorespiratory fitness (steps/minute) between baseline and immediate post-intervention (16 weeks).
Weight maintenance (Percent Body Fat) | 16 weeks
  Weight maintenance is defined as a change in % body fat less than ± 3% of baseline.
Weight maintenance (Body Mass Index) | 16 weeks
  Weight maintenance is defined as a change in body mass index (kg/m2) less than ± 3% of baseline.
Weight maintenance (Waist Circumference) | 16 weeks
  Weight maintenance is defined as a change in waist circumference less than ± 3% of baseline.
Change from baseline Moderate-to-vigorous physical activity (MVPA) | 40 weeks
  Minutes per week of MVPA is assessed a baseline and 24 weeks post-intervention (40 weeks) using accelerometry. The amount of change between baseline and 24 weeks post-intervention will be used to determine if the behavior was maintained.
Weight maintenance (Waist Circumference) | 40 weeks
  Weight maintenance is defined as a change in waist circumference less than ± 3% of baseline.
Weight maintenance (Body Mass Index) | 40 weeks
  Weight maintenance is defined as a change in body mass index (kg/m2) less than ± 3% of baseline.
Change from baseline in Physical Fitness | 40 weeks
  The 2-minute step in place test will be used to assess cardiorespiratory fitness (steps/minute).
Weight maintenance (Percent Body Fat) | 40 weeks
  Weight maintenance is defined as a change in % body fat less than ± 3% of baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Parra-Medina, PhD, Principal Investigator — UT Health San Antonio
Locations (1):
- University of Texas Health Science Center San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Salinas JJ, Parra-Medina D. Physical activity change after a promotora-led intervention in low-income Mexican American women residing in South Texas. BMC Public Health. 2019 Jun 20;19(1):782. doi: 10.1186/s12889-019-7105-6. PMID 31221117
- See also: Institute for Health Promotion Research Website — https://ihpr.uthscsa.edu/project/14